CLINICAL TRIAL: NCT02681263
Title: Efficacy of Temocillin in Urinary Tract Infection Due to ESBL Producing and AmpC Hyperproducing Enterobacteriaceae
Acronym: TEMO-ESBL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: French National Network of Clinical Research in Infectious Diseases (RENARCI) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC15.213; 2015-004178-14 (EudraCT Number)
Record Dates: First submitted 2015-11-27; First posted 2016-02-12 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — temocillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temocillin (Experimental): Treatment duration with a minimum of 5 days administration of the study drug: Temocillin (Negaban®) 6g/day (2g/tid) and as monotherapy.
  Total antibiotic treatment between 10 and 14 days according to local guidelines (up to 21 days in immunosuppressed patients).
  Interventions: Drug: Temocillin

INTERVENTIONS:
Drug: Temocillin — Treatment duration with a minimum of 5 days administration of the study drug: Temocillin (Negaban®) 6g/day (2g/tid) and as monotherapy.
  Other Names: NEGABAN

SUMMARY:
The present study aims at demonstrating the efficacy of temocillin in the treatment of UTI requiring parenteral therapy due to a confirmed ESBL producing or AmpC hyperproducing Enterobacteriaceae, resistant to quinolones and Bactrim® in France. In addition, this study will describe and support the use of high dose (6g/day) of temocillin which could be of interest for the treatment urinary tract infection due to multi-resistant bacteria having high MIC (up to 32 mg/L). The investigators will also evaluate the tolerance of the drug by monitoring the adverse event and the incidence of eventual Clostridium difficile associated infection.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 year old
* Patient benefits from social security
* Signed informed consent
* A urinary tract infection due to a confirmed ESBL producing strain (detected by the use of a rapid diagnostic test applied on the urine) requiring parenteral antimicrobial therapy
* Hospitalized patient
* For women able to procreate: Use of an acceptable method of birth control throughout the study. Acceptable methods of birth control are: oral contraceptives, intrauterine device (IUD), diaphragm with spermicide and condom. (All forms of hormonal contraception are acceptable

Exclusion Criteria:

* Patient infected with a bacteria which is not an ESBL-producing or AmpC hyperproducing Enterobacteriaceae
* Patients infected with a strain sensible to both fluoroquinolones and trimethoprim/sulfamethoxazole
* Patients infected with a strain resistant to temocillin
* Hospital-acquired urinary tract infection (defined as a urinary infection that occurred at least 48h post admission in the hospital)
* Patients has received any dose of active antimicrobial therapy (an antibiotic to which the infecting bacterium is susceptible) in the last 48h (prior to enrolment) except ≤ 2 dose of gentamicin.
* Patients presenting another site of infection than urinary (except onset of bacteraemia from urinary tract origin) due to Gram negative bacteria.
* Patients needing concomitant antimicrobial therapy.
* Septic shock
* Children (up to 18 years old)
* Women who is pregnant, breastfeeding, or expecting to conceive at any time during the study (pregnancy test will be conducted for woman without menopause)
* Patients with any kind of urinary/bladder catheter (JJ ureteral probe, …)
* Hypersensitivity to the active substance, to penicillins or to any other type of beta-lactam agent
* Chronically dialyzed patients
* Patients having a creatinine clearance < 30 mL/min
* Complete obstruction of the urinary tract
* Perinephretic or intrarenal abscesses
* Tutorship or curatorship patient
* Patient unable to give his consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Microbiological efficacy at Test of Cure in patients microbiologically evaluable | 7 days post end of Temocillin Treatment
  The microbiological efficacy will be assessed by quantitative urine culture and defined as follows:
  * Eradication : < 10^3 CFU/mL of the baseline pathogen
  * Persistence : ≥ 10^3 CFU/ml of the baseline pathogen
  * Superinfection : ≥ 10^5 CFU/ml of another uropathogen during therapy
  * New infection : ≥ 10^5 CFU/ml of another uropathogen after therapy
  * Relapse : eradication at TOC but ≥ 10^3 CFU/mL of the baseline pathogen at FU Overall microbiological response will be determined as "unfavorable" if persistence or superinfection or new infection or relapse.

SECONDARY OUTCOMES:
Clinical efficacy in clinical evaluable group | 3 weeks for end of Temocillin Treatment
  Each patient's response will be categorized as cure (resolution of all clinical symptoms), improvement (normalization of body temperature but persistence of either urinary syndrome or flank pain) or failure (persistence of baseline clinical symptoms or emergence of new symptoms related to UTI).
Microbiological efficacy | 3 weeks for end of Temocillin Treatment
  The microbiological efficacy will be assessed by quantitative urine culture and defined as follows:
  * Eradication : < 10^3 CFU/mL of the baseline pathogen
  * Persistence : ≥ 10^3 CFU/ml of the baseline pathogen
  * Superinfection : ≥ 10^5 CFU/ml of another uropathogen during therapy
  * New infection : ≥ 10^5 CFU/ml of another uropathogen after therapy
  * Relapse : eradication at TOC but ≥ 10^3 CFU/mL of the baseline pathogen at FU
Development of resistance to temocillin during treatment | 3 weeks for end of Temocillin Treatment
  The acquisition of resistance will be monitored in the central laboratory and is defined as an increase in MIC of at least 4 dilutions.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul STAHL, PU-PH, Study Chair — University Hospital, Grenoble
Locations (19):
- France (19):
  - CH Ajaccio, Ajaccio
  - CH Annecy Genevois, Annecy
  - APHP - Avicenne Hospital, Bobigny
  - APHP - Beaujon Hospital, Clichy
  - CHU de Martinique, Fort de France
  - CHU de Grenoble, Grenoble
  - APHP - Bicêtre Hospital, Le Kremlin-Bicêtre
  - CHU de Lille, Lille
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - APHP - Bichat Hospital, Paris
  - APHP - Cochin Hospital, Paris
  - APHP - St Louis, Paris
  - CH de Perpignan, Perpignan
  - CHU de Pointe à Pitre, Pointe à Pitre
  - CHU de Poitiers, Poitiers
  - CHU de Rouen, Rouen
  - CHU de Saint Etienne, Saint-Etienne
  - CHU de Tours, Tours

REFERENCES:
- [Background] Laterre PF, Wittebole X, Van de Velde S, Muller AE, Mouton JW, Carryn S, Tulkens PM, Dugernier T. Temocillin (6 g daily) in critically ill patients: continuous infusion versus three times daily administration. J Antimicrob Chemother. 2015 Mar;70(3):891-8. doi: 10.1093/jac/dku465. Epub 2014 Nov 27. PMID 25433006
- [Background] Balakrishnan I, Awad-El-Kariem FM, Aali A, Kumari P, Mulla R, Tan B, Brudney D, Ladenheim D, Ghazy A, Khan I, Virgincar N, Iyer S, Carryn S, Van de Velde S. Temocillin use in England: clinical and microbiological efficacies in infections caused by extended-spectrum and/or derepressed AmpC beta-lactamase-producing Enterobacteriaceae. J Antimicrob Chemother. 2011 Nov;66(11):2628-31. doi: 10.1093/jac/dkr317. Epub 2011 Aug 2. PMID 21810837
- [Background] Fournier D, Chirouze C, Leroy J, Cholley P, Talon D, Plesiat P, Bertrand X. Alternatives to carbapenems in ESBL-producing Escherichia coli infections. Med Mal Infect. 2013 Feb;43(2):62-6. doi: 10.1016/j.medmal.2013.01.006. Epub 2013 Feb 19. PMID 23433608
- [Background] Schulze B, Heilmann HD. Treatment of severe infections with temocillin. Clinical and bacteriological evaluation. Drugs. 1985;29 Suppl 5:207-9. doi: 10.2165/00003495-198500295-00046. PMID 4029026
- [Background] De Jongh R, Hens R, Basma V, Mouton JW, Tulkens PM, Carryn S. Continuous versus intermittent infusion of temocillin, a directed spectrum penicillin for intensive care patients with nosocomial pneumonia: stability, compatibility, population pharmacokinetic studies and breakpoint selection. J Antimicrob Chemother. 2008 Feb;61(2):382-8. doi: 10.1093/jac/dkm467. Epub 2007 Dec 10. PMID 18070831